CLINICAL TRIAL: NCT00565604
Title: Safety and Efficacy of Endovenous Laser Ablation for the Resolution of Incompetent Perforator Veins The RELIEVE Study
Brief Title: Safety and Efficacy of Endovenous Laser Ablation for the Resolution of Incompetent Perforator Veins
Acronym: RELIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Solutions LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0107; Protocol CP1002
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2011-03-17 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Venous Insufficiency
Keywords: Perforator Veins; Incompetent Veins; Varicose Veins
MeSH Terms: conditions — Venous Insufficiency; Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Short Catheter Delviery (Experimental): Patients with duplex ultrasound documented incompetent perforator veins will be treated using a short catheter delivery system in conjunction with a Bright Tip Laser fiber.
  Interventions: Device: Short Catheter Delivery

INTERVENTIONS:
Device: Short Catheter Delivery — For treating incompetent perforator veins of the lower extremities
  Other Names: Short Catheter 42-0664-01

SUMMARY:
This trial is designed as a prospective, non randomized, single center clinical trial to determine the safety and efficacy of laser ablation of incompetent perforator veins.

Within this clinical evaluation, fifty (50) limbs will be treated with Vari-Lase ®. A duplex ultrasound will verify the presence or absence of incompetent perforator veins (IPV). In addition, the number, diameter and location of the IPVs will be determined. Limbs with IPVs which measure greater than or equal to 3mm in diameter and are located superior to the foot and distal ankle will be considered for entry into the study.

DETAILED DESCRIPTION:
This is a non randomized, single center clinical investigation, evaluating a total of fifty (50) limbs for the treatment of venous stasis ulcerations using the Vari-Lase laser.

Subjects can be pre-screened utilizing standard of care data for the specified inclusion/exclusion criteria to ensure that they are eligible for treatment in the investigation. All subjects will have a mapping duplex ultrasound study in an Intersocietal Commission for the Accreditation of Vascular Laboratories (ICAVL) approved vascular laboratory. The ultrasound will verify the presence or absence of IPVs. The number, diameter, and location of the IPVs will be mapped. If the subject appears to qualify for the investigation, the subject will then be asked to give his/her written informed consent and be enrolled in the investigation. Upon satisfying all of the inclusion/exclusion criteria the subject will be accepted into the study.

After enrollment, the investigator will document the CEAP class, venous clinical severity score (VCSS), and venous disability score (VDS) in the subject's chart/medical record/source documentation for later transcription on the appropriate case report form. Digital photographs will be taken of the limb to be treated prior to treatment with the subject standing, following a standardized photography regimen.

All enrolled study participants will have a limb treated with the Vari-Lase laser manufactured by VSI. Subject preparation will be the same as for standard greater saphenous vein (GSV) or short saphenous vein, endovenous laser treatment. The initial technical success or failure of the procedure will be noted for each IPV and the pre-diameter of the IPV recorded. Multiple perforators may be treated in a single patient, as well as bilateral procedures allowed.

Follow-up duplex exams will be conducted within the first week of treatment and at 6 months. Follow-up duplex will verify patency vs. closure of IPV, and presence or absence of deep vein thrombosis (DVT) associated with that IPV. The goal is to prove successful closure of the treated IPVs veins as demonstrated by the duplex ultrasound at 6 weeks and show maintained closure of IPVs at 6 months.

Clinical examinations will occur at 2 weeks with an Associated Research Nurse Practitioner, at 6 weeks with the Medical Doctor, and at 6 months with either the Nurse Practitioner or Medical Doctor. At the 6 week visit, photos will be taken of the limb treated and there will be a reclassification of CEAP class, VDS, and VCSS.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years of age or older.
2. The subject has the presence of incompetent perforator veins measuring > 3 mm in diameter resultant of reflux documented on duplex ultrasound.
3. The subject has a CEAP classification of 3, 4, 5 or 6.
4. The subject has incompetent perforator veins that are superior to the foot and distal ankle.
5. The subject is willing and able to provide appropriate informed consent.
6. The subject is willing and able to comply with the requirements of the study protocol, including the predefined follow-up evaluations.

Exclusion Criteria:

1. The subject has a history of significant arterial disease.
2. The subject is known to be, or suspected to be, pregnant (verified in a manner consistent with institution's standard of care), or is lactating.
3. The subject has an Ankle Brachial Index (ABI) of < 0.5
4. The subject has occlusive thrombosis in the vein segment to be treated.
5. The subject has acute deep vein thrombosis.
6. The subject has an active or systemic infection.
7. The subject is or was enrolled in another investigational device or drug trial that may interfere with the results of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pepper, MD, Principal Investigator — Lake Washington Vascular Surgery
Locations (1):
- Lake Washington Vascular Surgery, Bellevue, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who had the presence of incompetent perforator veins were recruited from a medical clinic.
Pre-assignment Details: Two subjects were withdrawn from the study immediately after the index procedure due to failure to treat any incompetent perforator veins.
Groups:
- Short Catheter Delivery: Patients with duplex ultrasound documented incompetent perforator veins will be treated using a short catheter delivery system in conjunction with a Bright Tip Laser fiber.
Period: Overall Study
Arm/Group | Short Catheter Delivery
Started | 43
7 Day | 41
2 Week | 41
6 Week | 39
6 Month | 39
Completed | 39
Not Completed | 4
Not completed — Failure to treat | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Short Catheter Delivery
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Objective
Description: The primary objective is to demonstrate the clinical effectiveness (as determined by the absence of flow within the treated incompetent perforated vein [IPV])) of endovenous laser ablation. The number of treated IPVs that are closed at 6 weeks and remain closed at 6 months.
Time Frame: 6 Months
Population: The number of patients still participating in the study at 6-months.
Measure: Number; unit: Treated IPVs
Units Other Than Participants: Treated IPVs
Arm/Group | Short Catheter Delivery
Number analyzed (Participants) | 39
Number analyzed (Treated IPVs) | 76
Treated IPVs
  IPV Closure-6 months | 53
  IPV Closure-6 weeks | 66

2. Primary Outcome: Primary Safety Objective
Description: Safety: Evaluation of occurrence of major device-related adverse events through 6 weeks and the total at 6 months.
Time Frame: 6 Months
Population: The number of patients that were enrolled in the study.
Measure: Number; unit: Participants
Arm/Group | Short Catheter Delivery
Number analyzed (Participants) | 43
Participants
  Major Device-Related Adverse Events through 6 week | 14
  Major Device-Related Adverse Events Total 6 months | 15

3. Secondary Outcome: Secondary Effectiveness Objective
Description: Effectiveness: The reduction in patient symptoms and the satisfaction of the patient. Patient symptom assessment - CEAP Class, best=0 (no visible or palpable signs of venous disease) & worst=6 (Skin changes in conjunction with active ulceration), VDS, best=0 (asymptomatic) & worst=3 (unable to carry out usual activities even with compression and/or limb elevation) and VCSS, best=0 (absent) & worst=3 (severe). Patient satisfaction - modified Odom's criteria, best=excellent (I am very satisfied with the results of my laser treatment) & worst=poor (I am not satisfied with the results).
Time Frame: 6 Months
Population: The number of patients still participating in the study at 6-months.
Measure: Number; unit: Participants
Arm/Group | Short Catheter Delivery
Number analyzed (Participants) | 39
Participants
  CEAP Class Improved | 29
  VCSS Improved | 27
  VDS Improved | 30
  Patient Satisfaction (Good or Excellent) | 34

4. Secondary Outcome: Secondary Safety Objective
Description: Safety: Incidence rate of device-related minor adverse events.
Time Frame: 6 Months
Population: The number of subjects that were enrolled in the trial.
Measure: Number; unit: Participants
Arm/Group | Short Catheter Delivery
Number analyzed (Participants) | 43
Participants | 5

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subjects were assessed for adverse events at 1-week, 2-week, 6-week and 6-month follow-up office visits
Arm/Group | Short Catheter Delivery
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 15/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Catheter Delivery (N=43)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 6 (6)
Paresthesia (Nervous system disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less